CLINICAL TRIAL: NCT01655381
Title: A Multicenter, Open-label, Single Arm, Long-term Extension Study of WA19926 to Describe Safety During Treatment With Tocilizumab in Patients With Early, Moderate to Severe Rheumatoid Arthritis
Brief Title: A Long-Term Extension Study of WA19926 on the Safety of Tocilizumab (RoActemra/Actemra) in Participants With Early Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28174; 2011-005516-29 (EudraCT Number)
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (1):
- Tocilizumab (Experimental): Tocilizumab 8 milligrams per kilogram (mg/kg) administered intravenously once every 4 weeks during a minimum of 104 weeks.
  Interventions: Drug: Tocilizumab

INTERVENTIONS:
Drug: Tocilizumab — Tocilizumab 8 mg/kg administered intravenously.
  Other Names: RoActemra®; Actemra®

SUMMARY:
This open-label, single arm, multicenter long-term extension study will evaluate the safety and efficacy of tocilizumab (RoActemra/Actemra) in participants with moderate to severe rheumatoid arthritis who have completed the 104-week WA19926 core study. Eligible participants will receive tocilizumab 8 mg/kg intravenously every 4 weeks for up to 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult participants, >/= 18 years of age
* Participants who complete their last WA19926 core study visit (Week 104) and who may benefit from study drug treatment, at baseline or later if they are in remission DAS28 at Week 104 of WA19926, according to the Investigator's assessment
* No current or recent adverse event or laboratory finding preventing the use of the study drug dose of tocilizumab 8 mg/kg at baseline visit
* Women of childbearing potential must agree to use adequate contraception as defined by protocol during and up to 3 months after treatment

Exclusion Criteria:

* Pregnant females
* Participants who have withdrawn prematurely from the WA19926 core study for any reason
* Treatment with any investigational agent or cell-depleting therapies since the last administration of study drug in WA19926
* Treatment with an anti-tumor necrosis factor (TNF) or anti-interleukin (IL) 1 agent, or a T-cell costimulation modulator since the last administration of study drug in WA19926
* Immunization with a live/attenuated vaccine since the last administration of study drug in WA19926
* Diagnosis since last WA19926 visit (Week 104) of rheumatic autoimmune disease other than rheumatoid arthritis
* Diagnosis since last WA19926 visit (Week 104) of inflammatory joint disease other than rheumatoid arthritis
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies, including tocilizumab and its excipients
* Evidence of severe uncontrolled concomitant disease or disorder
* Known active or history of recurrent infections
* Active tuberculosis requiring treatment in the previous 3 years
* History of alcohol, drug or chemical abuse since inclusion in the WA19926 study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- France (6):
  - Cahors
  - Montpellier
  - Mulhouse
  - Orléans
  - Paris
  - Toulouse

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total 15 participants who completed the Week 104 visit of the WA19926 core study, were enrolled in this follow-up open-label extension study.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 15
Completed | 12
Not Completed | 3
Not completed — Investigator Decision | 1
Not completed — Moved to Another City | 1
Not completed — Insufficient Treatment Response | 1

BASELINE CHARACTERISTICS:
Population: Analysis was performed in Included population, defined as all participants who entered the study.
Groups:
- Tocilizumab: Tocilizumab 8 mg/kg administered intravenously once every 4 weeks during a minimum of 104 weeks.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (9.1)
Gender [Count of Participants; unit: Participants]
  Female | 12
  Male | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Any Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) is any AE that is fatal; life-threatening; requires or prolongs inpatient hospitalization; results in persistent or significant disability/incapacity; congenital anomaly/birth defect in a neonate/infant or significant medical event in the Investigator's judgment. AE of special interest (AESI) includes serious and/or medically significant infectious; myocardial infarction(MI) / acute coronary syndrome (ACS); gastrointestinal (GI) perforation; anaphylaxis / hypersensitivity reactions; demyelinating disorders; stroke; serious and/or medically significant bleeding events; serious and/or medically significant hepatic events; malignancies malignant.
Time Frame: Up to 160 weeks
Population: Safety population is defined as all included participants who received having at least one tocilizumab administration.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
percentage of participants
  AE | 93.3
  SAE | 6.7
  Non-serious AE | 93.3
  Tocilizumab-related AE | 80.0
  Tocilizumab-related SAE | 0
  Tocilizumab-related non-SAE | 80.0
  AESI | 20.0
  Tocilizumab-related AESI | 20.0
  AE leading to dose modification | 33.3
  AE leading to Tocilizumab discontinuation | 6.7
  AE leading to death | 0

2. Secondary Outcome: Percentage of Participants With at Least One Clinical Remission Period
Description: Clinical remission: Disease Activity Score Based on 28-joint Count and Erythrocyte Sedimentation Rate (DAS28-ESR) less than (<)2.6 and/or Simplified Disease Activity Index (SDAI) less than or equal to (≤)3.3 for a period of at least two consecutive assessment visits (every 12 weeks) over the extension study period. DAS28-ESR was calculated using Swollen Joint Count Based on 28 Joints (SJC28), Tender Joint Count Based on 28 Joints (TJC28), ESR (mm/hour) and patient's global assessment of disease activity (100-millimeter (mm) horizontal visual analog scale with 0=no disease activity to 100=maximum disease activity. DAS28-ESR scores range from 0-10, with higher scores corresponding to greater disease activity. SDAI was calculated using SJC28, TJC28, C-reactive protein (CRP) (milligrams per liter (mg/L)), the patient's global assessment of disease activity and physician's global assessment of disease activity; SDAI scores range from 0-86, where lower scores indicate less disease activity.
Time Frame: Up to approximately 148 weeks
Population: The included population includes all participants who entered the study. All included participants were part of safety population.
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
percentage of participants | 100.0

3. Secondary Outcome: Percentage of Participants With at Least One Drug-Free Period
Description: Drug-free remission period was defined as clinical remission for at least 2 consecutive assessment visits (every 12 weeks) AND without tocilizumab administration during this clinical remission period.
Time Frame: Up to approximately 148 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
percentage of participants | 13.3

4. Secondary Outcome: Cumulative Time of Remission Per Participant Over the Extension Study Period
Description: Clinical remission was defined as DAS28-ESR <2.6 and/or SDAI ≤3.3 for a period of at least two consecutive assessment visits (every 12 weeks) over the extension study period. DAS28-ESR scores range from 0 to 10, with higher scores corresponding to greater disease activity. SDAI scores range from 0 to 86, where lower scores indicate less disease activity.
Time Frame: Up to approximately 148 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
days | 598.00 [179.0 to 1,072.0]

5. Secondary Outcome: Percentage of Participants With at Least 1 Rheumatoid Arthritis (RA) Flare
Description: An RA flare was defined as an increase in DAS28-ESR from the previous available visits of >1.2, or >0.6 if current DAS28-ESR ≥3.2. DAS28-ESR scores range from 0 to 10, with higher scores corresponding to greater disease activity.
Time Frame: Up to approximately 148 weeks
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
percentage of participants | 40.0

6. Secondary Outcome: Time to RA Flare Following Remission or Drug-Free Remission
Description: Time to RA flare was defined as period of clinical remission or drug-free remission followed by flare of DAS28-ESR (increase in DAS28-ESR from the previous available visits of >1.2, or >0.6 if current DAS28-ESR ≥3.2). In the case of several remission periods for the same participant, the largest period was used.
Time Frame: Up to approximately 148 weeks
Population: as for outcome 2
Measure: Median (Full Range); unit: days
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
days | 289.0 [179.0 to 739.0]

7. Secondary Outcome: Change From Day 1 in DAS28-ESR Scores Over Time
Description: DAS28-ESR was calculated using Swollen Joint Count Based on 28 Joints (SJC28), Tender Joint Count Based on 28 Joints (TJC28), ESR (mm/hour) and patient's global assessment of disease activity (100-millimeter (mm) horizontal visual analog scale with 0=no disease activity to 100=maximum disease activity. DAS28-ESR scores range from 0 to 10, with higher scores corresponding to greater disease activity.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: The included population includes all participants who entered the study. All included participants were part of safety population. Here, n = number of participants who were evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
units on a scale
  Day 1 (n = 14) | 2.09 (1.12)
  Change at Week 12 (n = 10) | -0.43 (0.96)
  Change at Week 24 (n = 13) | -0.65 (1.86)
  Change at Week 36 (n = 11) | -0.03 (1.42)
  Change at Week 48 (n = 13) | -0.58 (1.46)
  Change at Week 56 (n = 11) | -1.02 (1.50)
  Change at Week 68 (n = 11) | -1.39 (1.31)
  Change at Week 80 (n = 10) | -0.83 (1.33)
  Change at Week 92 (n = 10) | -0.69 (1.50)
  Change at Week 104 (n = 10) | -0.94 (1.44)
  Change at Week 116 (n = 6) | -1.15 (1.37)
  Change at Week 128 (n = 2) | 0.40 (1.70)
  Change at Week 140 (n = 1) | 0.10 (NA) — Standard deviation was not estimable as 1 participant was evaluated.

8. Secondary Outcome: Change From Day 1 in Simplified Disease Activity Index (SDAI) Scores Over Time
Description: SDAI was calculated using SJC28, TJC28, C-reactive protein (CRP) (milligrams per liter (mg/L)), and the patient's global assessment of disease activity and physician's global assessment of disease activity; SDAI scores range from 0 to 86, where lower scores indicate less disease activity.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
units on a scale
  Day 1 (n = 6) | 4.40 (3.67)
  Change at Week 12 (n = 6) | -1.70 (3.43)
  Change at Week 24 (n = 4 | 2.68 (17.12)
  Change at Week 36 (n = 0) | NA (NA) — Mean and standard deviation was not estimable as no participants was evaluated.
  Change at Week 48 (n = 3) | -3.70 (3.21)
  Change at Week 56 (n = 3) | -2.90 (1.64)
  Change at Week 68 (n = 2) | -7.30 (3.54)
  Change at Week 80 (n = 3) | -3.37 (3.42)
  Change at Week 92 (n = 4) | -2.05 (5.11)
  Change at Week 104 (n = 2) | -6.10 (0.14)
  Change at Week 116 (n = 3) | -4.77 (2.46)
  Change at Week 128 (n = 0) | NA (NA) — Mean and standard deviation was not estimable as no participants was evaluated.
  Change at Week 140 (n = 1) | -0.90 (NA) — Standard deviation was not estimable as 1 participant was evaluated.

9. Secondary Outcome: Change From Day 1 in Tender Joint Count Based on 28 Joints (TJC28) Over Time
Description: The number of tender joints was recorded on the joint assessment form at each visit, no tenderness = 0, tenderness = 1; total was calculated by adding all the joints for a maximum score of 28 tender joints. Higher scores correspond to greater disease activity.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: tender joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
tender joints
  Day 1 (n = 15) | 2.07 (5.62)
  Change at Week 12 (n = 15) | -0.87 (6.58)
  Change at Week 24 (n = 14) | 0.29 (9.22)
  Change at Week 36 (n = 14) | 1.00 (8.68)
  Change at Week 48 (n = 14) | 1.07 (9.24)
  Change at Week 56 (n = 13) | -1.77 (6.26)
  Change at Week 68 (n = 12) | -1.42 (5.92)
  Change at Week 80 (n = 11) | -2.45 (6.67)
  Change at Week 92 (n = 12) | -0.67 (3.75)
  Change at Week 104 (n = 11) | -1.82 (7.05)
  Change at Week 116 (n = 6) | -1.00 (0.89)
  Change at Week 128 (n = 3) | 0.67 (2.08)
  Change at Week 140 (n = 1) | -1.00 (NA) — Standard deviation was not estimable as 1 participant was evaluated.

10. Secondary Outcome: Change From Day 1 in Swollen Joint Count Based on 28 Joints (SJC28) Over Time
Description: The number of swollen joints was recorded on the joint assessment form at each visit, no swelling = 0, swelling =1; total was calculated by adding all the joints for a maximum score of 28 swollen joints. Higher scores correspond to greater disease activity.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Mean (Standard Deviation); unit: swollen joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
swollen joints
  Day 1 (n = 15) | 0.33 (0.62)
  Change at Week 12 (n = 15) | 0.27 (1.44)
  Change at Week 24 (n = 14) | 0.50 (2.03)
  Change at Week 36 (n = 14) | 1.50 (2.71)
  Chnage at Week 48 (n = 14) | 0.29 (1.38)
  Change at Week 56 (n = 13) | 0.46 (2.07)
  Change at Week 68 (n = 12) | -0.08 (1.16)
  Change at Week 80 (n = 11) | 0.09 (1.38)
  Change at Week 92 (n = 12) | 0.50 (2.35)
  Change at Week 104 (n = 11) | 0.55 (1.86)
  Change at Week 116 (n = 6) | -0.17 (1.72)
  Change at Week 128 (n = 3) | 0.00 (0.00)
  Change at Week 140 (n = 1) | 0.00 (NA) — Standard deviation was not estimable as 1 participant was evaluated.

11. Secondary Outcome: Erythrocyte Sedimentation Rate (ESR) Over Time
Description: ESR is an direct measure of how much inflammation is in the body. The normal range is 0-22 mm/hour for men and 0-29 mm/hour for women. Higher scores correspond to greater disease activity.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Median (Full Range); unit: mm/hour
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
mm/hour
  Day 1 (n = 14) | 10.0 [1.0 to 61.0]
  Week 12 (n = 11) | 2.00 [1.0 to 20.0]
  Week 24 (n = 14) | 2.50 [1.0 to 24.0]
  Week 36 (n = 12) | 2.00 [1.0 to 26.0]
  Week 48 (n = 14) | 2.00 [1.0 to 19.0]
  Week 56 (n = 13) | 2.00 [1.0 to 9.0]
  Week 68 (n = 12) | 2.50 [1.0 to 13.0]
  Week 80 (n = 11) | 3.00 [2.0 to 6.0]
  Week 92 (n = 11) | 2.00 [1.0 to 20.0]
  Week 104 (n = 11) | 2.00 [1.0 to 30.0]
  Week 116 (n= 6) | 2.00 [2.0 to 15.0]
  Week 128 (n= 3) | 3.00 [2.0 to 4.0]
  Week 140 (n= 1) | 10.00 [10.0 to 10.0]

12. Secondary Outcome: C-reactive Protein (CRP) Level
Description: C-reactive protein (CRP) is a blood test marker for inflammation in the body. Normal CRP levels are below 5 milligrams per liter (mg/L). Higher scores correspond to greater disease activity.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Median (Full Range); unit: mg/L
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
mg/L
  Day 1 (n = 6) | 4.70 [0.5 to 24.0]
  Week 12 (n = 11) | 2.00 [0.3 to 10.0]
  Week 24 (n = 11) | 2.00 [0.2 to 9.0]
  Week 36 (n = 6) | 0.85 [0.3 to 2.0]
  Week 48 (n = 8) | 1.30 [0.2 to 5.0]
  Week 56 (n = 9) | 2.00 [0.2 to 21.0]
  Week 68 (n = 7) | 2.00 [0.5 to 12.0]
  Week 80 (n = 8) | 2.00 [0.3 to 10.7]
  Week 92 (n = 8) | 2.00 [0.3 to 25.0]
  Week 104 (n = 7) | 2.00 [0.3 to 22.5]
  Week 116 (n= 4) | 2.00 [2.0 to 3.0]
  Week 128 (n= 1) | 2.00 [2.0 to 2.0]
  Week 140 (n= 1) | 4.00 [4.0 to 4.0]

13. Secondary Outcome: Participants' Global Assessment of Pain (VAS) Score
Description: The participants' global assessment of pain (VAS) was assessed using a 100-mm horizontal VAS with 0=no pain to 100=maximum pain.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
units on a scale
  Day 1 (n = 15) | 11.00 [0.0 to 50.0]
  Week 12 (n = 15) | 7.00 [0.0 to 37.0]
  Week 24 (n = 14) | 9.00 [0.0 to 75.0]
  Week 36 (n = 14) | 10.00 [0.0 to 66.0]
  Week 48 (n = 14) | 8.00 [0.0 to 64.0]
  Week 56 (n = 13) | 4.00 [0.0 to 50.0]
  Week 68 (n = 12) | 4.00 [0.0 to 25.0]
  Week 80 (n = 11) | 19.00 [1.0 to 40.0]
  Week 92 (n = 12) | 8.50 [0.0 to 50.0]
  Week 104 (n = 11) | 9.00 [0.0 to 24.0]
  Week 116 (n= 6) | 3.50 [0.0 to 20.0]
  Week 128 (n= 3) | 3.00 [1.0 to 20.0]
  Week 140 (n= 1) | 6.00 [6.0 to 6.0]

14. Secondary Outcome: Participants' Global Assessment of Disease Activity (VAS) Score
Description: The participants' global assessment of disease activity (VAS) was assessed using a 100-mm horizontal VAS with 0=no disease activity to 100=maximum disease.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
units on a scale
  Day 1 (n = 15) | 13.00 [0.0 to 30.0]
  Week 12 (n = 15) | 17.00 [0.0 to 75.0]
  Week 24 (n = 14) | 18.50 [0.0 to 80.0]
  Week 36 (n = 14) | 10.00 [0.0 to 68.0]
  Week 48 (n = 14) | 7.50 [0.0 to 49.0]
  Week 56 (n = 13) | 5.00 [0.0 to 50.0]
  Week 68 (n = 12) | 5.00 [0.0 to 32.0]
  Week 80 (n = 11) | 24.00 [1.0 to 70.0]
  Week 92 (n = 12) | 10.50 [0.0 to 30.0]
  Week 104 (n = 11) | 10.00 [0.0 to 57.0]
  Week 116 (n= 6) | 4.00 [0.0 to 15.0]
  Week 128 (n= 3) | 7.00 [2.0 to 10.0]
  Week 140 (n= 1) | 15.00 [15.0 to 15.0]

15. Secondary Outcome: Physicians' Global Assessment of Disease Activity (VAS) Score
Description: The physicians' global assessment of disease activity (VAS) was assessed using a 100-mm horizontal VAS with 0=no disease activity to 100=maximum disease.
Time Frame: Day 1 and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
units on a scale
  Day 1 (n = 15) | 5.00 [0.0 to 20.0]
  Week 12 (n = 15) | 6.00 [0.0 to 21.0]
  Week 24 (n = 13) | 1.00 [0.0 to 60.0]
  Week 36 (n = 14) | 5.00 [0.0 to 55.0]
  Week 48 (n = 14) | 5.00 [0.0 to 50.0]
  Week 56 (n = 13) | 6.00 [0.0 to 60.0]
  Week 68 (n = 12) | 4.50 [0.0 to 13.0]
  Week 80 (n = 11) | 3.00 [0.0 to 18.0]
  Week 92 (n = 12) | 9.0 [0.0 to 43.0]
  Week 104 (n = 11) | 5.00 [0.0 to 40.0]
  Week 116 (n= 6) | 5.00 [0.0 to 10.0]
  Week 128 (n= 3) | 15.00 [1.0 to 30.0]
  Week 140 (n= 1) | 5.00 [5.0 to 5.0]

16. Secondary Outcome: Percentage of Participants With Health Assessment Questionnaire Disability Index (HAQ-DI) Remission
Description: HAQ-DI remission was defined as HAQ-DI score <0.5.
  HAQ-DI is the participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Baseline and Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128 140
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Groups:
- Tocilizumab: Tocilizumab 8 mg/kg administered intravenously once every 4 weeks through Week 104.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
percentage of participants
  Baseline (n = 15) | 73.3
  Week 12 (n = 9) | 66.7
  Week 24 (n = 8) | 62.5
  Week 36 (n = 10) | 60.0
  Week 48 (n = 10) | 50.0
  Week 56 (n = 10) | 60.0
  Week 68 (n = 9) | 77.8
  Week 80 (n = 9) | 66.7
  Week 92 (n = 8) | 75.0
  Week 104 (n = 7) | 71.4
  Week 116 (n= 3) | 100
  Week 128 (n= 1) | 100
  Week 140 (n= 1) | 100

17. Secondary Outcome: Percentage of Participants With Clinically Meaningful Improvement From Baseline in HAQ-DI
Description: Clinically meaningful improvement was defined as an improvement in HAQ-DI score of ≥0.22.
  HAQ-DI is the participant-reported assessment of ability to perform tasks in 8 categories of daily living activities: dress/groom; arise; eat; walk; reach; grip; hygiene; and common activities over past week. Each item scored on 4-point scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Overall score was computed as the sum of domain scores and divided by the number of domains answered. Total possible score range 0-3 where 0 = least difficulty and 3 = extreme difficulty.
Time Frame: Weeks 12, 24, 36, 48, 56, 68, 80, 92, 104, 116, 128, 140
Population: as for outcome 7
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 15
percentage of participants
  Week 12 (n = 9) | 33.3
  Week 24 (n = 8) | 25.0
  Week 36 (n = 10) | 40.0
  Week 48 (n = 10) | 30.0
  Week 56 (n = 10) | 30.0
  Week 68 (n = 9) | 33.3
  Week 80 (n = 9) | 22.2
  Week 92 (n = 8) | 12.5
  Week 104 (n = 7) | 28.6
  Week 116 (n= 3) | 100
  Week 128 (n= 1) | 100
  Week 140 (n= 1) | 100

ADVERSE EVENTS:
Time Frame: Up to 160 weeks
Description: An adverse event was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Safety population, defined as all included participants having at least one tocilizumab administration.
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 1/15
Other Adverse Events (participants affected / at risk) | 14/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=15)
Oedema peripheral (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=15)
Bronchitis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 2
Pharyngitis (Infections and infestations) | 2
Tracheitis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 2
Ear infection (Infections and infestations) | 1
Fungal infection (Infections and infestations) | 1
Gingivitis (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Periodontitis (Infections and infestations) | 1
Pertussis (Infections and infestations) | 1
Rhinitis (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tooth abscess (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Vulvovaginal mycotic infection (Infections and infestations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Tendon pain (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Asthenia (General disorders) | 4
Chest pain (General disorders) | 1
Fatigue (General disorders) | 1
Inflammatory pain (General disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Intertrigo (Skin and subcutaneous tissue disorders) | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Alanine aminotransferase increased (Investigations) | 1
Colonoscopy (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Interferon gamma release assay positive (Investigations) | 1
Transaminases increased (Investigations) | 1
Weight decreased (Investigations) | 1
Insomnia (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Abdominal pain (Gastrointestinal disorders) | 1
Anal fissure (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Limb injury (Injury, poisoning and procedural complications) | 2
Tooth avulsion (Injury, poisoning and procedural complications) | 1
Tooth fracture (Injury, poisoning and procedural complications) | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2
Decreased appetite (Metabolism and nutrition disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 2
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Cataract operation (Surgical and medical procedures) | 1
Dental cleaning (Surgical and medical procedures) | 1
Eye laser surgery (Surgical and medical procedures) | 1
Joint injection (Surgical and medical procedures) | 1
Tooth extraction (Surgical and medical procedures) | 1
Tympanic membrane disorder (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Eyelid oedema (Eye disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Allergy to arthropod bite (Immune system disorders) | 1
Radicular pain (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.